CLINICAL TRIAL: NCT00724919
Title: Association of Antibiotic Utilization Measures and Control of Extended-Spectrum β-Lactamases (ESBLs) (A Post-Intervention Surveillance Study)
Brief Title: A Post-Intervention Surveillance Study Regarding the Acquisition Rate of ESBL-KP, Ecoli
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Other Study IDs: 0910X-101440
Record Dates: First submitted 2008-07-23; First posted 2008-07-30 (Estimated); Last update posted 2008-08-11 (Estimated); Status verified 2008-08

CONDITIONS: Infection
Keywords: ESBL
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
To determine the acquisition rate of ESBL producing E. coli or K. pneumoniae, post- intervention in the selected medical centres

DETAILED DESCRIPTION:
This is post-interventional study to follow the acquisition rate of ESBP producing E. coli or K. pneumoniae at the sites involved in a previous interventional study.

ELIGIBILITY:
Inclusion

1. All patients admitted or transferred to ICU/burn unit.
2. Patients of either sex, 18 years of age or older. Exclusion

Patients were excluded if they had underlying conditions or diseases that were ultimately fatal within 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to ICU/burn unit
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2003-12; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
The acquisition rate of ESBL producing E. coli or K. pneumoniae at the end of surveillance phase | 48hours

SECONDARY OUTCOMES:
The infection rate due to ESBL producing E. coli, or due to K. pneumoniae at the end of surveillance phase | 48hours

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (2):
- Taiwan (2):
  - Miaoli County
  - Taichung